CLINICAL TRIAL: NCT04421157
Title: The Effectiveness of Two Different Exercises in Adolescent Idiopathic Scoliosis: A Single-blind Study
Brief Title: Exercises in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Hikmet Kocaman, Research Assistant, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaramanogluMehmetbeyU
Record Dates: First submitted 2020-05-12; First posted 2020-06-09 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis, Scoliosis, Exercise
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Each patient selected a number in a closed envelope, which was sorted via the 'Research Randomiser' program for the randomisation process, and the patients were separated into the following two groups; Schroth group (n=14) and stabilization group (n=14)
Who Masked: Outcomes Assessor
Masking Description: Assessments were undertaken at baseline, and after the 10 week treatment period for each patient by the investigator, who was blind to the allocation of the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth group (Experimental): The Schroth group received Schroth exercises in addition to traditional rehabilitation.
  Interventions: Other: Schroth Exercises
- Stabilization group (Experimental): The stabilization group received core stabilization in addition to traditional rehabilitation.
  Interventions: Other: Core stabilization Exercises

INTERVENTIONS:
Other: Schroth Exercises — The Schroth approach consists of 3D scoliosis-specific exercises based on kinesthetic and sensorimotor principles. The goal of Schroth exercises is to teach patients to consciously maintain the correct posture in daily living activities in order to improve the curve, pain, and self-image. The treatment program consists of scoliotic posture correction and a breathing pattern with the help of proprioceptive and exteroceptive stimulations and mirror control. Traditional exercises program included strengthening back, abdominal, pelvis and shoulder girdle muscles and also muscles in the convex side of the curve, stretching exercises especially for the concave side of the curve, postural training, flexibility exercises for the spine, and breathing exercises. Schroth group received Schroth exercises in addition to traditional rehabilitation for 10 weeks. Patients received 30 sessions for 90 minutes at the clinic for ten-week treatment period.
  Other Names: Schroth Method; Scoliosis specific exercises
  Arms: Schroth group
Other: Core stabilization Exercises — Each exercise session consisted of a warm-up exercise, core stabilization exercise, and a cool-down exercise. The core stabilization exercise was designed with consideration of local, global muscle stability training, global muscle mobility training,and strengthening training of these core structures was carried out progressively advancing more difficult. Traditional exercises program included strengthening back, abdominal, pelvis and shoulder girdle muscles and also muscles in the convex side of the curve, stretching exercises especially for the concave side of the curve, postural training, flexibility exercises for the spine, and breathing exercises. The Stabilization group received Core stabilization in addition to traditional rehabilitation for 10 weeks. Patients received 30 sessions for 90 minutes at the clinic for ten-week treatment period.
  Arms: Stabilization group

SUMMARY:
The purpose of this study was to investigate the effectiveness of two different exercises in adolescent idiopathic scoliosis. In total, 28 subjects with adolescent idiopathic scoliosis were randomly divided into two groups: Schroth (n = 14) and stabilization group (n = 14). The Schroth group received Schroth exercises in addition to traditional rehabilitation, and the stabilization group received core stabilization in addition to traditional rehabilitation for 10 weeks. The outcome measures were based on Cobb angle, angle of trunk rotation, spinal mobility, cosmetic trunk deformity, muscle strength, and quality of life.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a progressive growth disease with unknown etiology, characterized by a three-dimensional deformity of the spine (frontal translation, sagittal modification, and torsion of the spinous processes on the concave side of the scoliotic curve on radiographs).

In patients with AIS, in addition to curve progression there are many problems commonly occur such as; muscular imbalance, functional limitations, altered posture, gait deviations, reduced flexibility of the spine, back pain, negative physico-social, body image effects, and in severe cases pulmonary symptoms. The asymmetry of the trunk and pelvis are affected related to the shape and angle of scoliosis, and the weight distribution position changes depending on the shape and the Cobb angle of scoliosis. To deal with these complications and more, various treatment approaches have been proposed for AIS, including exercise, bracing, casting, traction, biofeedback, surgery, and simple observation to prevent, correct or halt the progression of the deformity. Conservative treatment methods including physiotherapy and bracing are accepted in Central Europe.

In literature, exercises are recommended to decrease progression, to improve spine and thoracic cage flexibility, muscle strengths, and elasticity, to correct postural behavior, and neuro-motor control, spine stability. In general, traditional exercises (TE) including postural training, stretching, and strengthening exercises for spinal musculature, respiratory exercises have been used for many years for scoliosis. Except for the traditional exercises, there are several exercise concepts including Schroth, Side Shift, Dobomed methods... etc. Schroth exercises are asymmetric scoliosis-specific postural exercises that aim to improve the curve, function, posture, self-image, and pain. Schroth exercises target strength and endurance training of the back, abdominal, and leg muscles. Also one of the aim of Schroth exercises is to improve motor control of the posture by repeating corrective movements with progressively less feedback. Schroth exercises are the most studied scoliosis exercises but there are limited randomized controlled studies on Schroth exercises.

Recently general physiotherapeutic exercises including, Core stabilization (CS) exercises, Pilates have been used in the conservative treatment of idiopathic scoliosis. CS exercises are described as therapy techniques that improve postural control, and functional stability through increasing neuromuscular control, the strength of trunk stabilization muscles, the endurance of postural muscles around the spine, the balance between pelvis and spine. However, limited studies are determining CS exercises' effect on patients with AIS. In a study CS exercises found to be more effective in reducing pain and rotational deformity than traditional exercises in the conservative rehabilitation of AIS.

A recent systematic review showed that therapeutic exercise had been effective to reduce symptoms, Cobb's angle, trunk rotation, craniovertebral angle, and body asymmetries, and to improve muscular endurance, pulmonary function, and functional capacity of patients with AIS. Corrective, therapeutic exercises appear to have positive effects by improving function and reducing symptoms, as well as various angles and body asymmetries. However, further studies with better methodological quality are required to confirm these outcomes and detect the best therapeutic exercise intervention. And also there is a need for randomized controlled studies on different methods of exercise to choose the most effective exercise in clinical practice.

There was no research compared to the effects of the Schroth method and CS exercises in patients with AIS. And also there was no research examining the effects of the Schroth method on peripheral muscle strengths. This study aimed to investigate the effects of the Schroth versus CS exercises in addition to traditional exercises, on Cobb angle, trunk rotation, peripheral muscle strengths, spine mobility, cosmetic deformity, and health-related quality of life in patients with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of adolescent idiopathic scoliosis,
* A Cobb angle of 10 to 30 degrees
* Having Lenke type 1 curve
* No other treatment which might affect scoliosis

Exclusion Criteria:

* Non-idiopathic scoliosis
* Prescribed brace
* Surgical correction history
* Who were unable to participate in the supervised sessions,or those who refused to follow treatment were excluded.
* Contraindications to exercise -Accompanying mental problems, neurological- muscular or rheumatic diseases,

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Cobb's angle | 10 week
  Cobb's angles were measured on standard standing anterior-posterior spine radiograph and recorded as degrees. Cobb angle is considered the gold standard to evaluate the curve magnitude. The Cobb angle is the angle from a posterior-anterior full spine radiographs between the upper endplate of the upper-end vertebra of the largest curve and the lower endplate of the lower end vertebra from the largest curve.

SECONDARY OUTCOMES:
Trunk rotation angles | 10 week
  -Trunk rotation angles Axial trunk rotations (ATR) were assessed with a scoliometer in Adam's forward bend test.
Muscle strength | 10 week
  Muscle strengths were assessed by a Biodex System 4-Pro dynamometer (Biodex, Inc., Shirley, New York). Upper extremity pattern strengths (flexion-abduction-external rotation / extension-adduction-internal rotation), and quadriceps, hamstring muscles strengths were assessed in both extremity. The outcome parameter was the peak torque (expressed in Nm) which was normalized to the participants' body weight (expressed in Nm/kg) in an effort to reduce inter-subject variability in raw scores of quantitative muscle tests.
Spinal mobility | 10 week
  Spinal mobility was assessed with a new computer-aided skin-surface device (The Spinal Mouse® System, Idiag, Fehraltorf, Switzerland). Spinal Mouse is an external non-invasive measurement method developed to evaluate the motility and shape of the spine in many planes. The Spinal Mouse has acceptable metrological properties to assess segmental and global thoracal and lumbar mobility. Measurements were performed between spinous process of C7 and the top of the anal crease (approximately S3). Maximal extension, maximal flexion and maximal left and right lateral flexion positions were performed. The analysis of spinal mobility in the sagittal (SAP - maximal extension to flexion) and the coronal (CRP - maximal left to right flexion) plane was evaluated.
Cosmetic trunk deformity | 10 week
  Walter Reed Visual Assessment Scale (WRVAS) was used to assess cosmetic deformity. The domains of WRVAS are body curve, rib prominence, flank prominence, head rib pelvis, head pelvis, shoulder level, and scapular rotation. Each domain generates a score from 1 (best deformity) to 5 (worst deformity). The total score is an average of these 7 domains.
SRS-22 Questionnaire | 10 week
  The SRS-22 questionnaire assesses the quality of life in scoliosis. It is a self-reported tools assessing self-image, function, pain, mental health with 5 questions each and satisfaction with care with 2 questions which are scored from 1 (best answer) to 5 (worst answer) each question. A total score is based on all 22 questions and an average of these 7 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Hikmet Kocaman, MSc, Principal Investigator — Karamanoğlu Mehmetbey University
Locations (1):
- Karamanoglu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romano M, Minozzi S, Zaina F, Saltikov JB, Chockalingam N, Kotwicki T, Hennes AM, Negrini S. Exercises for adolescent idiopathic scoliosis: a Cochrane systematic review. Spine (Phila Pa 1976). 2013 Jun 15;38(14):E883-93. doi: 10.1097/BRS.0b013e31829459f8. PMID 23558442
- [Background] Shneerson JM, Madgwick R. The effect of physical training on exercise ability in adolescent idiopathic scoliosis. Acta Orthop Scand. 1979 Jun;50(3):303-6. doi: 10.3109/17453677908989771. PMID 474101
- [Background] Negrini S, Fusco C, Minozzi S, Atanasio S, Zaina F, Romano M. Exercises reduce the progression rate of adolescent idiopathic scoliosis: results of a comprehensive systematic review of the literature. Disabil Rehabil. 2008;30(10):772-85. doi: 10.1080/09638280801889568. PMID 18432435
- [Background] Schreiber S, Parent EC, Khodayari Moez E, Hedden DM, Hill DL, Moreau M, Lou E, Watkins EM, Southon SC. Schroth Physiotherapeutic Scoliosis-Specific Exercises Added to the Standard of Care Lead to Better Cobb Angle Outcomes in Adolescents with Idiopathic Scoliosis - an Assessor and Statistician Blinded Randomized Controlled Trial. PLoS One. 2016 Dec 29;11(12):e0168746. doi: 10.1371/journal.pone.0168746. eCollection 2016. PMID 28033399
- [Background] Schreiber S, Parent EC, Hill DL, Hedden DM, Moreau MJ, Southon SC. Patients with adolescent idiopathic scoliosis perceive positive improvements regardless of change in the Cobb angle - Results from a randomized controlled trial comparing a 6-month Schroth intervention added to standard care and standard care alone. SOSORT 2018 Award winner. BMC Musculoskelet Disord. 2019 Jul 8;20(1):319. doi: 10.1186/s12891-019-2695-9. PMID 31286903
- [Background] Thompson JY, Williamson EM, Williams MA, Heine PJ, Lamb SE; ACTIvATeS Study Group. Effectiveness of scoliosis-specific exercises for adolescent idiopathic scoliosis compared with other non-surgical interventions: a systematic review and meta-analysis. Physiotherapy. 2019 Jun;105(2):214-234. doi: 10.1016/j.physio.2018.10.004. Epub 2018 Oct 27. PMID 30824243
- [Background] Ceballos Laita L, Tejedor Cubillo C, Mingo Gomez T, Jimenez Del Barrio S. Effects of corrective, therapeutic exercise techniques on adolescent idiopathic scoliosis. A systematic review. Arch Argent Pediatr. 2018 Aug 1;116(4):e582-e589. doi: 10.5546/aap.2018.eng.e582. English, Spanish. PMID 30016036
- [Background] Kim G, HwangBo PN. Effects of Schroth and Pilates exercises on the Cobb angle and weight distribution of patients with scoliosis. J Phys Ther Sci. 2016 Mar;28(3):1012-5. doi: 10.1589/jpts.28.1012. Epub 2016 Mar 31. PMID 27134403
- [Background] Nault ML, Allard P, Hinse S, Le Blanc R, Caron O, Labelle H, Sadeghi H. Relations between standing stability and body posture parameters in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1911-7. doi: 10.1097/00007632-200209010-00018. PMID 12221357
- [Background] Sanders JO, Polly DW Jr, Cats-Baril W, Jones J, Lenke LG, O'Brien MF, Stephens Richards B, Sucato DJ; AIS Section of the Spinal Deformity Study Group. Analysis of patient and parent assessment of deformity in idiopathic scoliosis using the Walter Reed Visual Assessment Scale. Spine (Phila Pa 1976). 2003 Sep 15;28(18):2158-63. doi: 10.1097/01.BRS.0000084629.97042.0B. PMID 14501929
- [Background] Coelho DM, Bonagamba GH, Oliveira AS. Scoliometer measurements of patients with idiopathic scoliosis. Braz J Phys Ther. 2013 Mar-Apr;17(2):179-84. doi: 10.1590/S1413-35552012005000081. PMID 23778766
- [Background] Alves de Araujo ME, Bezerra da Silva E, Bragade Mello D, Cader SA, Shiguemi Inoue Salgado A, Dantas EH. The effectiveness of the Pilates method: reducing the degree of non-structural scoliosis, and improving flexibility and pain in female college students. J Bodyw Mov Ther. 2012 Apr;16(2):191-8. doi: 10.1016/j.jbmt.2011.04.002. Epub 2012 Jan 5. PMID 22464116
- [Background] Martinez-Llorens J, Ramirez M, Colomina MJ, Bago J, Molina A, Caceres E, Gea J. Muscle dysfunction and exercise limitation in adolescent idiopathic scoliosis. Eur Respir J. 2010 Aug;36(2):393-400. doi: 10.1183/09031936.00025509. Epub 2009 Dec 23. PMID 20032022
- [Background] Gur G, Ayhan C, Yakut Y. The effectiveness of core stabilization exercise in adolescent idiopathic scoliosis: A randomized controlled trial. Prosthet Orthot Int. 2017 Jun;41(3):303-310. doi: 10.1177/0309364616664151. Epub 2016 Sep 13. PMID 27625122
- [Background] Ameer MA, Kamel MI, Elhafez YM. A comparison of sagittal spine deformities among elementary school students using spinal mouse device. Work. 2019;64(3):545-550. doi: 10.3233/WOR-193015. PMID 31658087
- [Background] Livanelioglu A, Kaya F, Nabiyev V, Demirkiran G, Firat T. The validity and reliability of "Spinal Mouse" assessment of spinal curvatures in the frontal plane in pediatric adolescent idiopathic thoraco-lumbar curves. Eur Spine J. 2016 Feb;25(2):476-82. doi: 10.1007/s00586-015-3945-7. Epub 2015 Apr 22. PMID 25900295
- [Background] Cheshire J, Gardner A, Berryman F, Pynsent P. Do the SRS-22 self-image and mental health domain scores reflect the degree of asymmetry of the back in adolescent idiopathic scoliosis? Scoliosis Spinal Disord. 2017 Dec 11;12:37. doi: 10.1186/s13013-017-0144-9. eCollection 2017. PMID 29238754
- [Background] Tsai YT, Leong CP, Huang YC, Kuo SH, Wang HC, Yeh HC, Lau YC. The electromyographic responses of paraspinal muscles during isokinetic exercise in adolescents with idiopathic scoliosis with a Cobb's angle less than fifty degrees. Chang Gung Med J. 2010 Sep-Oct;33(5):540-50. PMID 20979705
- [Background] Lin JJ, Chen WH, Chen PQ, Tsauo JY. Alteration in shoulder kinematics and associated muscle activity in people with idiopathic scoliosis. Spine (Phila Pa 1976). 2010 May 15;35(11):1151-7. doi: 10.1097/BRS.0b013e3181cd5923. PMID 20421854
- [Derived] Kocaman H, Bek N, Kaya MH, Buyukturan B, Yetis M, Buyukturan O. The effectiveness of two different exercise approaches in adolescent idiopathic scoliosis: A single-blind, randomized-controlled trial. PLoS One. 2021 Apr 15;16(4):e0249492. doi: 10.1371/journal.pone.0249492. eCollection 2021. PMID 33857180